CLINICAL TRIAL: NCT02878343
Title: A Randomized Controlled Trial of Incentives Versus Environmental Strategies for Weight Loss
Brief Title: The Healthy Weigh Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 821428
Record Dates: First submitted 2016-07-25; First posted 2016-08-25 (Estimated); Results first posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Fertility

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Incentives (Active Comparator): Daily lottery type incentives tied to achievement of weight loss goals
  Interventions: Behavioral: Incentives
- Environmental strategies (Active Comparator): Individually tailored environmental strategies around food intake and physical activity; automated text/emails sent from study website platform
  Interventions: Behavioral: Environmental strategies
- Incentive and environmental strategies (Active Comparator): A combination of incentives and environmental strategies
  Interventions: Behavioral: Incentives; Behavioral: Environmental strategies
- Usual care (No Intervention): Standard employee wellness benefits

INTERVENTIONS:
Behavioral: Incentives — Daily lottery type incentives tied to achievement of weight loss goals
  Arms: Incentive and environmental strategies; Incentives
Behavioral: Environmental strategies — Individually tailored environmental strategies around food intake and physical activity; automated text/emails sent from study website platform
  Arms: Environmental strategies; Incentive and environmental strategies

SUMMARY:
This study will evaluate the comparative effectiveness of behavioral economic financial incentives and environmental strategies, separately and together, in achieving initial weight loss and maintenance of weight loss, in obese employee populations. Our study contributes to the Centers for Disease Control and Prevention's efforts to combat obesity but in particular to the Centers for Disease Control's winnable battles (physical activity and obesity); the National Center for Chronic Disease Prevention and Health Promotion's strategic priorities around well-being, health equity, and evaluation and dissemination of environmental and systems-wide solutions to address public health problems; and the National Center for Chronic Disease Prevention and Health Promotion's domain around healthier work-site initiatives, the Centers for Disease Control and Prevention's efforts to improve nutrition and physical activity to prevent obesity, and reduction of cardiovascular disease risk. This study is a 4-arm randomized controlled trial in which 344 employees of the City of Philadelphia, Independence Blue Cross, and South Eastern Pennsylvania Transportation Authority with initial Body Mass Index of 30 will be randomized to receive one of the following: 1) Daily lottery type incentives tied to achievement of weight loss goals (incentive arm); 2) individually tailored environmental strategies around food intake and physical activity (environmental arm); 3) a combination of incentives and environmental strategies (combined arm); or 4) standard employee wellness benefits and weigh-ins every 6 months (control arm). Phase I of the study (first 6 months) will focus on weight loss; Phase II (months 7-18) will focus on continued weight loss or maintenance for those who choose to maintain weight loss as opposed to continuing to try to lose weight; Phase III (months 19-24) will provide a period of post-intervention follow-up to measure sustainability of effects.

DETAILED DESCRIPTION:
Analysis Plan 11.1 Statistical Considerations Descriptive analyses We will produce data summaries regularly using frequencies for categorical variables and means, medians, and ranges for continuous variables. We will assess data quality and examine distributional assumptions with graphical methods. To evaluate balance among groups achieved by randomization, we will compare baseline values of all variables across the 4 arms using appropriate tests.

General procedures All primary analyses will be on an intent-to-treat basis including each participant in the group to which s/he was randomized, regardless of adherence to the assigned strategy. Given the high rates of missing data typical of weight loss studies, handling of missing data is an important issue. Primary analyses will use multiple imputation for the missing in-person weight outcome at 18 months, using the randomization strata (sex, employer, initial BMI), study arm and other baseline variables as predictors in the imputation model. Baseline variables will include age, race, income, education, marital status, household size, physical activities, eating behavior index, stages of change, SF-36 General Health, and baseline weight. Sensitivity analyses will be performed with imputation models that also use post-baseline data, , and recent weight loss trend before drop out, as well as an analysis that assumes that any participants for whom follow-up weight loss data are unavailable have had their weight return to baseline (weight at beginning of Pre Phase). Within each arm, this last assumption is likely to be conservative but this may not be the case in inter-arm comparisons, depending on the dropout rates in the different arms and true follow-up weights of the dropouts. Thus, a key secondary analysis will consider the effect of differential dropout among the treatment arms. For this analysis, methods that address potential patterns of MNAR may be considered in the missing data imputation, such as pattern mixture models as appropriate. Finally, we will also consider a per-protocol type analysis, which examines the difference in the intervention arms in the complete case data.

Efficacy Analyses All hypotheses will be tested using two-sided, 0.05-level tests unless otherwise specified (notably the Holm testing approach will be used for the five primary hypotheses in Specific Aims 1-4). The primary analyses will be an unadjusted intent-to-treat analyses, using a t-test for differences in weight change from baseline to 18 months, as measured by the in-person weight, between each intervention group and the control group, and the combined compared to each single intervention, applying the Holm p-value correction for multiple comparisons testing. If weight change appears to be non-normally distributed in the blinded data, we will find an appropriate. Missing data will be handled as described above.

Weight change between baseline and 18 months, with 95% confidence intervals (CIs), will be estimated for comparison with adjusted analyses. We will estimate regression models adjusted for the stratification variables (sex, employer, initial BMI) and other participant characteristics factors including age, race, income, and education. We will evaluate the evidence of confounding for other baseline variables (baseline weight, marital status, household size, physical activities- i.e total minutes of MVPA+walking/week, eating behavior index, stages of change, SF-36 General Health) using change in estimate criterion (10%). We will fit exploratory models of the repeated weight measurements that incorporate time as a polynomial function or using visit-specific indicator variables to determine the most parsimonious model that adequately describes the observed patterns, as necessary. Models will be built separately for the in-person and at home weight data. Models using the at-home weight data would be considered only as potential exploratory analyses comparing the 3 intervention arms, since at-home weights are not available for the control arm. We will investigate random-effects models that allow for baseline individual variability as well as variability in the changes in weights over time; an example is the following: E(weightij) = ß0 +ß1Timej + ß2Groupi+ ß3Xi + b0i + b1i Timej, where i indicates subject, j indicates assessment times, the parameters are fixed effects linking time, a treatment group vector, and a vector of other demographic or clinical covariates Xi to the outcomes, and b0i and b1i are random intercept and slope effects. Tests for significance of random effects will use likelihood ratio tests for nested models; we will compare models with different random effects structures using the maximized log-likelihoods and the Akaike Information Criterion (AIC). We will apply standard diagnostic techniques to assess model adequacy. We will use treatment by time interactions to assess whether the rate of change in weight differs by intervention arm. We hypothesize that incentives may be more effective among lower income individuals and will evaluate this using interaction terms of income with treatment group. We will explore differential effects by race and education and baseline levels of intrinsic motivation and stages of change. We will also consider other potential mediators, such as the home food and activity environment. To assess the sensitivity of treatment effect estimates to missing data, we mayfit hierarchical or mixed effects models with and without accounting for informative missing data.

For Specific Aim 5, we will consider appropriate methods for cost effective analysis such as the models proposed below. We will assess the costs of each of the intervention arms from both the employer and social perspective and compare the cost differences between each arm relative to the effectiveness measured by incremental weight loss achieved. The principal incremental cost-effectiveness ratios between intervention and control arms will be from the employer's perspective and we will compare costs during the intervention from baseline to 18 months per unit change in weight. Secondary analyses may also 1) evaluate this same ratio but use either 6 months post- intervention data (24 month visit) or 12 months of intervention data (12 month visit) and 2) evaluate these 2 ratios using a limited social perspective. Cost models will use a generalized linear model with a log link and gamma family. Missing data strategies will parallel those described above. We will assess sampling uncertainty for the comparison of costs and effects by calculating parametric 95% CIs for the cost per kg lost and acceptability curves. Standard errors and correlation of the difference in cost and effect will be derived using a bootstrap procedure.

11.2 Power and Sample Size Considerations We have designed the study with adequate power to detect differences in weight loss over an 18-month period. Our intervention should achieve its maximal impact in maintaining initial weight loss at the end of Phase II (month 18), when the incentive payments cease. To maintain the experiment-wide Type I error and guard against false conclusions of effectiveness, we will use the Holm multiple comparisons adjustment for test the 5 primary comparisons in Specific Aims 1-4 . If the interventions are as effective as hypothesized, the proposed sample size maintains greater than 90% power to show significance for each of the three intervention arms compared to control and greater than 80% power to show significance for the combined intervention group compared to each of the two interventions alone.

It is important to note that while we originally planned to recruit 328 participants, a small subset was unable to successfully set up their Withings scales post randomization due to Wi-Fi connectivity issues. Therefore, we increased our target sample size by the number of people who were unable to connect their Withings scales to the Way To Health platform (16 additional subjects), bringing our recruitment total to 344 participants. The final statistical analysis is adjusted for the stratification factors to account for any imbalances that may have occurred. We have previously communicated this information to the IRB and the members of the Data Safety and Monitoring Board (DSMB), who approved this approach. The following information outlines our original power calculations and sample size considerations.

We plan to recruit approximately one third of the participants required for the start of Phase I from each of our participating employers (IBC, SEPTA, and City of Philadelphia). Given the large number of potentially eligible employees, we can, if needed, easily increase the proportion of participants from any of these employers to meet recruitment targets. Participants will be randomized to our 3 intervention groups and the control group using a 1:1 ratio for the intervention arms. We built in a margin of 20% of our original target sample size of 328 for potential attrition before the 18-month assessment, resulting in an expected 260 participants (65 per arm) who are available for analysis at the end of Phase II. This sample size will provide us with greater than 90% power to detect a difference in weight change between baseline and the 18-month weigh-in of 5 kg between each single intervention group and the control group (primary outcomes for Specific Aims 1-3) and 87% power to detect a 3 kg difference between the combined group and either the incentive or environmental strategies groups (Specific Aim 4). Namely, we will have greater than 85% power for the 5 primary comparisons of interest for an expected weight change between months 0-18 of -8 kg, -5 kg and 0 kg in the combined, intervention and control groups, respectively (a net difference between single intervention and control groups of 5 kg, combined intervention and control groups of 8 kg, and 3kg between the single interventions and combined group) and assuming a standard deviation (S.D.) of weight loss of 5 kg. We will also have greater than 80% power to detect a difference of 4.6 kg in weight change between single intervention and control groups and 7.3 kg between the combined and control groups (primary outcomes for Specific Aims 1-3), while maintaining approximately 80% power for a 2.7 kg difference between the combined and each single intervention (Specific Aim 4). For our secondary outcomes (Specific Aim 5), we wish to compare the cost differences between each arm relative to the effectiveness measured by incremental weight loss achieved. We will calculate a point estimate of cost per kg of weight loss based on estimated inter-arm differences in weight loss and the incremental cost of the interventions, as described in C.3.d.ii.c. For weight loss at 18 months, given an expected incremental cost of $810 (incentives) and incremental weight loss of 5 kg, 328 participants provide 80% power to detect a cost per kg lost of $430 and greater than 90% power to detect a cost per kg lost of $575. This study is primarily a test of the efficacy of these interventions. Due to resource constraints and because we do not yet know about intervention effectiveness, we did not power this study based on cost effectiveness analyses. Estimated detectable costs per kg are a function of wide confidence intervals due to sample size.

11.3 Measurement of effect: The goal of this analysis will be to assess relative weight loss in the intervention arms relative to control. For the principal cost-effectiveness analysis, measurement of incremental weight loss will be based on differences in weight between baseline and the 18 month visit; in secondary analyses it will be based on weight differences between baseline and 24 months and baseline and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Men and women > 18 yrs. of age
* Full-time or part-time employees at Southeastern Pennsylvania Transportation Authority , Independence Blue Cross, or the City of Philadelphia
* BMI of 30 to 55 kg/m2
* Participants must receive their health benefits from Independence Blue Cross; one of our partners in the study

Exclusion Criteria:

* Unstable heart disease, uncontrolled hypertension, kidney disease, and other serious chronic illness (e.g., transplant recipient, terminal illness)
* Substance abuse; bulimia nervosa or related behaviors; or diabetes medication other than metformin
* Pregnancy or breast feeding
* Contraindications to counseling about diet, physical activity, or weight reduction
* Unstable mental illness
* Individuals unable to read consent forms or fill out surveys in English will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 344 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Volpp, MD, PhD, Principal Investigator — The University of Pennsylvania; Karen Glanz, PhD, MPH, Principal Investigator — The University of Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Glanz K, Kather C, Chung A, Choi JR, Volpp KG, Clapp J. Qualitative study of perceptions of factors contributing to success or failure among participants in a US weight loss trial of financial incentives and environmental change strategies. BMJ Open. 2024 Mar 29;14(3):e078111. doi: 10.1136/bmjopen-2023-078111. PMID 38553057
- [Derived] Glanz K, Shaw PA, Kwong PL, Choi JR, Chung A, Zhu J, Huang QE, Hoffer K, Volpp KG. Effect of Financial Incentives and Environmental Strategies on Weight Loss in the Healthy Weigh Study: A Randomized Clinical Trial. JAMA Netw Open. 2021 Sep 1;4(9):e2124132. doi: 10.1001/jamanetworkopen.2021.24132. PMID 34491350

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Incentives | Environmental Strategies | Incentive and Environmental Strategies | Usual Care
Started | 86 | 86 | 86 | 86
Completed | 65 | 66 | 65 | 66
Not Completed | 21 | 20 | 21 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Incentives | Environmental Strategies | Incentive and Environmental Strategies | Usual Care | Total
Number analyzed (Participants) | 86 | 86 | 86 | 86 | 344
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 86 | 86 | 86 | 86 | 344
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.4 (9.5) | 46.6 (10.9) | 44.9 (11.1) | 44.6 (10.6) | 45.6 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 61 | 61 | 64 | 247
  Male | 25 | 25 | 25 | 22 | 97
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 37 | 43 | 49 | 43 | 172
  White | 38 | 35 | 30 | 35 | 138
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 11 | 8 | 7 | 8 | 34
Region of Enrollment [Number; unit: participants]
  United States | 86 | 86 | 86 | 86 | 344

OUTCOME MEASURES:

1. Primary Outcome: Mean Weight Change
Description: Change in mean weight (lbs.) from baseline to 18 months
Time Frame: Baseline to 18 months
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Incentives | Environmental Strategies | Incentive and Environmental Strategies | Usual Care
Number analyzed (Participants) | 86 | 86 | 86 | 86
pounds | -6.86 (2.30) | -6.86 (2.08) | -2.82 (1.94) | -0.66 (1.69)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the 18 month study period.
Description: Definition does not differ from ct.gov definitions.
Arm/Group | Incentives | Environmental Strategies | Incentive and Environmental Strategies | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/86 | 0/86 | 0/86 | 0/86
Serious Adverse Events (participants affected / at risk) | 2/86 | 1/86 | 1/86 | 1/86
Other Adverse Events (participants affected / at risk) | 0/86 | 0/86 | 0/86 | 0/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Incentives (N=86) | Environmental Strategies (N=86) | Incentive and Environmental Strategies (N=86) | Usual Care (N=86)
Aortic valve replacement (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Diagnostic tests showed enlarged heart, leakage from aortic valve, and a hole in his heart. Aortic valve replacement/repair of hole in heart on 10/1/15. Good reports on 2 post-op checkups. Prescribed 2-3 months of cardiac rehab.
Vehicular accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 — Involved in a vehicular accident, fractured C 3,4,5 vertebrae; surgery on 8/10/15 w/placement of titanium plates and a soft cast. Two post-op appointments; cleared and no recommended rehab.
Headaches and dizziness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Subject had recurring headaches with some episodes of dizziness upon standing. MRI revealed white lesions on brain, caused by HBP. Originally diagnosed with HBP in 7/2015 & on Clonidine. BP was normal range at last 2 visits to PCP.
Heart attack (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Heart attack, admitted on 8/15, discharged on 8/20; cardiac therapy protocol at Penn Presby., returned to work 10/15
Brain hemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Admitted to ER, tests reveal brain hemorrhage; cause unknown. Had 2 seizures while in transport to ER. Emergency surgery to release pressure on the brain, w/successful outcome. Prescribed 2yr. regimen of Keppra.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-06-26): https://cdn.clinicaltrials.gov/large-docs/43/NCT02878343/Prot_SAP_000.pdf
  • Informed Consent Form (2015-08-01): https://cdn.clinicaltrials.gov/large-docs/43/NCT02878343/ICF_001.pdf